CLINICAL TRIAL: NCT06492681
Title: Correlation Between Optic Nerve Sheath Diameter Measured by POCUS and Neurological Deficit in Physical Examination in Adult Patients With Suspected Ischemic Stroke Evaluated in Emergency Departments
Brief Title: Correlation Between Optic Nerve Sheath Diameter and Neurological Deficit in Adult Patients With Suspected Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Clinica Mexico (Other)
Responsible Party: Principal Investigator, Jose Ivan Rodriguez de Molina Serrano, Head of Research and Critical Care Medicine, Clinica Mexico
Other Study IDs: 00001
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
Keywords: optic nerve sheath diameter; stroke; emergency department
MeSH Terms: conditions — Ischemic Stroke; Stroke; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The ultrasound of the optic nerve sheath diameter (ONSD) is a non-invasive tool used in the detection of intracranial hypertension and other neurological conditions. The aim of this research is to evaluate the correlation between the ultrasound measurement of the optic nerve sheath diameter and the side of neurological focus in the physical examination of adult patients evaluated in emergency departments.

DETAILED DESCRIPTION:
II. Hypothesis The ultrasound measurement of the optic nerve sheath diameter correlates with the side of neurological focus in the physical examination of adult patients evaluated in emergency departments.

III. Objectives Estimate the correlation between the ultrasound measurement of the optic nerve sheath diameter and the side of neurological focus in the physical examination of adult patients evaluated in emergency departments.

Determine the sensitivity and specificity of the ultrasound measurement of the optic nerve sheath diameter for predicting the side of neurological focus.

IV. Methodology

Study design:

A observational study will be conducted in a secondary care hospital.

Population and sample:

Adult patients (≥18 years) presenting to the emergency department with neurological symptoms, such as headache, altered level of consciousness, motor or sensory deficit, among others, will be included. Patients with contraindications for ocular ultrasound or with a history of previous ocular surgery will be excluded.

Procedures:

1. Informed consent will be obtained from patients who meet the inclusion criteria.
2. A neurological physical examination will be performed to identify the side of neurological focus.
3. The optic nerve sheath diameter will be measured using ultrasound with a high-frequency linear transducer (7.5-12 MHz).
4. Demographic, clinical, and ultrasound data will be recorded for the patients.

Data analysis:

The correlation between the ultrasound measurement of the optic nerve sheath diameter and the side of neurological focus will be calculated using Pearson's or Spearman's correlation coefficient, depending on the distribution of the data. Additionally, sensitivity, specificity, positive and negative predictive values, and 95% confidence intervals will be calculated to determine the diagnostic utility of the ultrasound measurement of the optic nerve sheath diameter in identifying the side of neurological focus.

V. Ethical considerations The ethical guidelines established by the Declaration of Helsinki will be followed, and the privacy and confidentiality of patients will be protected. The protocol will be approved by the hospital's Research Ethics Committee before its implementation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected acute ischemic stroke
* CT scan negative to hemorrhagic stroke
* Informed consent

Exclusion Criteria:

* Contraindications to perform ocular ultrasound
* Patients with ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to include a diverse adult population, encompassing various ages, genders, and ethnic backgrounds, reflective of the general demographic seen in emergency departments with suspected ischemic stroke. By doing so, the study seeks to enhance the generalizability of its findings across different subgroups within the adult population.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation between optic nerve sheath and side of clinical neurological focalization | In the first 4 hours of arrival to Emergency Department
  Estimate the correlation between the ultrasound measurement of the optic nerve sheath diameter and the side of neurological focus in the physical examination of adult patients evaluated in emergency departments.

SECONDARY OUTCOMES:
sensitivity and specificity of the ultrasound measurement of the optic nerve sheath diameter for predicting the side of neurological focus. | In the first 4 hours of arrival to Emergency Department
  Determine the sensitivity and specificity of the ultrasound measurement of the optic nerve sheath diameter for predicting the side of neurological focus.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Mexico, Piedras Negras, Coahuila, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lau T, Ahn JS, Manji R, Kim DJ. A Narrative Review of Point of Care Ultrasound Assessment of the Optic Nerve in Emergency Medicine. Life (Basel). 2023 Feb 15;13(2):531. doi: 10.3390/life13020531. PMID 36836888
- [Background] Nathani A, Ghamande SA, Kambhampati S, Anderson B, Lohse M, White HD. The Use of POCUS-Obtained Optic Nerve Sheath Diameter in Intracerebral Hemorrhage. POCUS J. 2023 Nov 27;8(2):170-174. doi: 10.24908/pocus.v8i2.16563. eCollection 2023. PMID 38099170
- [Background] Rajajee V, Vanaman M, Fletcher JJ, Jacobs TL. Optic nerve ultrasound for the detection of raised intracranial pressure. Neurocrit Care. 2011 Dec;15(3):506-15. doi: 10.1007/s12028-011-9606-8. PMID 21769456
- [Background] Bauerle J, Lochner P, Kaps M, Nedelmann M. Intra- and interobsever reliability of sonographic assessment of the optic nerve sheath diameter in healthy adults. J Neuroimaging. 2012 Jan;22(1):42-5. doi: 10.1111/j.1552-6569.2010.00546.x. Epub 2010 Dec 1. PMID 21121998
- [Background] Kimberly HH, Shah S, Marill K, Noble V. Correlation of optic nerve sheath diameter with direct measurement of intracranial pressure. Acad Emerg Med. 2008 Feb;15(2):201-4. doi: 10.1111/j.1553-2712.2007.00031.x. PMID 18275454